CLINICAL TRIAL: NCT00000161
Title: Randomized Trials of Vitamin Supplements and Eye Disease
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Eye Institute (NEI) (NIH)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: NEI-63
Record Dates: First submitted 1999-09-23; First posted 1999-09-24 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-09

CONDITIONS: Macular Degeneration; Cataract
Keywords: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration; Cataract | interventions — Aspirin; beta Carotene; Ascorbic Acid; Vitamin E

INTERVENTIONS:
Drug: Aspirin
Drug: Beta-Carotene
Drug: Vitamin C
Drug: Vitamin E

SUMMARY:
To determine whether vitamin E supplementation reduces the risk of cataract and age-related macular degeneration (AMD) in women.

To determine whether vitamin C supplementation reduces the risk of cataract and AMD in women.

To determine whether beta-carotene supplementation reduces the risk of cataract and AMD in women.

To determine whether alternate day, low-dose aspirin reduces the risk of cataract and AMD in women.

To identify potential risk factors for cataract and AMD including cigarette smoking, alcohol intake, blood pressure, blood cholesterol, cardiovascular disease, height, body mass index, and diabetes.

DETAILED DESCRIPTION:
Cataract and AMD are two of the most important causes of visual impairment in older Americans. Approximately 3.3 million people have visual impairment due to cataract. Cataract extraction, although one of the safest and most successful of all operations, is now the most frequently performed operation in the United States among persons older than 60, costing an estimated $1.5 billion annually. AMD is the leading cause of new cases of blindness in persons aged 65 and older. Approximately 25 percent of persons aged 65 years and older have signs of AMD. The pathogenesis of AMD, however, is only partly understood, and its etiology remains obscure. For most patients, there is no available treatment. The public health burden imposed by cataract and AMD will only increase in the coming decades as the U.S. population ages.

These randomized, double-masked, placebo-controlled trials will test the hypotheses that supplementation with antioxidant vitamins and with low-dose aspirin reduces the risk of age-related cataract and AMD. The study populations are the Women's Health Study (WHS) and the Women's Antioxidant Cardiovascular Study (WACS). The WHS is a randomized, double-masked, placebo-controlled trial using a 2x2 factorial design to test low-dose aspirin (100 mg on alternate days) and vitamin E (600 IU on alternate days) in the primary prevention of cardiovascular disease (CVD) and cancer. It is being conducted among 39,876 apparently healthy female health professionals age 45 years and older. The WACS is a randomized, double-masked, placebo-controlled secondary prevention trial using a 2x2x2x2 factorial design to test antioxidant vitamins (vitamins E [600 IU on alternate days] and C [500 mg daily], beta carotene [50 mg on alternate days]), and a combination of folate (800 mg daily), vitamin B6 (25 mg daily), and vitamin B12 (1 mg daily) among women who are at high risk for CVD morbidity and mortality. It is being conducted among 8,171 female health professionals, ages 40 years or older, who either have preexisting CVD or have at least three coronary risk factors and therefore are at high risk for the development of CVD.

In addition to the randomized comparisons, the investigators will also examine risk factors for age-related cataract and AMD in these two populations. Factors to be examined include cigarette smoking, alcohol intake, blood pressure, blood cholesterol, cardiovascular disease, height, body mass index, diabetes, and dietary factors.

In each study population, followup questionnaires were sent at 6 and 12 months after randomization and every 12 months thereafter requesting information about development of relevant study end points including cataract and AMD and participant compliance with study medications. Reported diagnoses of cataract and AMD are confirmed by medical record review. The primary analysis for the randomized studies will be incidence of AMD or cataract in the treatment and placebo groups. Survival analysis will be used to determine whether there is a difference in time to AMD or cataract diagnosis.

ELIGIBILITY:
Women's Health Study:

A participant must have met all of the following criteria:

(a) female; (b) aged 45 years or older; (c) postmenopausal or with no intention of becoming pregnant; (d) no reported personal history of cardiovascular disease, cancer (other than non-melanoma skin cancer), gout, peptic ulcer, chronic renal or liver disease, or other serious illness precluding participation; (e) no reported history of serious side effects to the study treatments; (f) not currently taking aspirin, aspirin containing medication, or nonsteroidal anti-inflammatory drugs (NSAIDs) more than 1 day per week or, if so doing, willing to forego use of these medications; (g) not currently taking individual supplements of vitamin E or beta carotene more than 1 day per week; (h) not currently taking anticoagulants or corticosteroids.

Women's Antioxidant Cardiovascular Study:

Potentially eligible female health professionals for WACS were identified from the pool of respondents to the Women's Health Study initial mailing and must have met the following criteria:

(a) female; (b) date of birth before January 1, 1955; (c) a reported history of myocardial infarction (MI), stroke (CVA), angina pectoris (AP), coronary artery bypass grafting (CABG), percutaneous transluminal angioplasty (PCTA), transient ischemic attack (TIA), carotid endarterectomy (CEA), or peripheral artery surgery (PAS); (d) no history of cancer (except non-melanoma skin cancer) within the past 10 years and no active liver disease or cirrhosis; (e) pregnancy physiologically impossible due to menopause (natural or surgical) or tubal ligation, or the participant does not intend to become pregnant in the future as indicated on the initial WHS questionnaire; (f) no current use of a vitamin K-depleting anticoagulant agent (e.g., Coumadin). Individuals taking aspirin or other NSAIDs were not excluded.

Min Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 1993-08

REFERENCES:
- [Derived] Christen WG, Glynn RJ, Chew EY, Albert CM, Manson JE. Folic acid, pyridoxine, and cyanocobalamin combination treatment and age-related macular degeneration in women: the Women's Antioxidant and Folic Acid Cardiovascular Study. Arch Intern Med. 2009 Feb 23;169(4):335-41. doi: 10.1001/archinternmed.2008.574. PMID 19237716